CLINICAL TRIAL: NCT06178367
Title: Effectiveness and Safety Comparison Between Moisturizers Containing Low Molecular Weight Hyaluronic Acid, High Molecular Weight Hyaluronic Acid, and Vehicle on Skin Hydration in the Elderly With Xerotic Skin
Brief Title: Effectiveness and Safety of Topical Hyaluronic Acid of Different Molecular Weights in Xerotic Skin Treatment
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Parikesit Muhammad, Dermatology and Venereology Resident, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 23061046
Record Dates: First submitted 2023-12-10; First posted 2023-12-21 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Xerosis Cutis

STUDY DESIGN:
Intervention Model Description: This is a split study, one participant receive three interventions in three area in the leg. The distribution of treatment groups is carried out randomly using the block randomization method.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All moisturizers used in this clinical trial were made in the same preparation and packaging
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Topical 0,1% low molecular weight (7 kDa) hyaluronic acid (Experimental): Participants receive moisturizer containing 0,1% low molecular weight (7 kDa) hyaluronic acid on 7 cm x 7 cm area on the right or left leg based on the randomization, twice a day for 1 month
  Interventions: Drug: Low molecular weight hyaluronic acid
- Topical 0,1% high molecular weight (1.800 kDa) hyaluronic acid (Active Comparator): Participants receive moisturizer containing 0,1% high molecular weight (1.800 kDa) hyaluronic acid on 7 cm x 7 cm area on the right or left leg based on the randomization, twice a day for 1 month
  Interventions: Drug: High molecular weight hyaluronic acid
- Vehicle (Placebo Comparator): Participants receive vehicle on 7 cm x 7 cm area on the right or left leg based on the randomization, twice a day for 1 month.
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: Low molecular weight hyaluronic acid — Topical 0,1% low molecular weight (7 kDa) hyaluronic acid in vehicle
  Other Names: LMWHA
  Arms: Topical 0,1% low molecular weight (7 kDa) hyaluronic acid
Drug: High molecular weight hyaluronic acid — Topical 0,1% high molecular weight (1.800 kDa) hyaluronic acid in vehicle
  Other Names: HMWHA
  Arms: Topical 0,1% high molecular weight (1.800 kDa) hyaluronic acid
Drug: Vehicle — Vehicle ingredients including aqua, paraffinum liquidum, glycerin, petrolatum, hydroxyethyl acrylate/sodium acryloyldimethyl taurate copolymer, arachidyl alcohol, squalane, behenyl alcohol, phenoxyethanol, arachidyl glucoside, allantoin, chlorphenesin, and disodium EDTA
  Other Names: Placebo
  Arms: Vehicle

SUMMARY:
The goal of this clinical trial is to compare 0,1% topical low molecular weight (7 kDa) hyaluronic acid with 0,1% high molecular weight (1.800 kDa) hyaluronic acid as therapy of xerotic skin in elderly

DETAILED DESCRIPTION:
This clinical trial is conducted to compare the effectiveness and safety between moisturizers containing 0,1% low molecular weight hyaluronic acid, 0,1% high molecular weight hyaluronic acid, and its vehicle on skin hydration of elderly with xerotic skin. It is designed to answer following questions:

1. Is the skin capacitance in the elderly after using moisturizers containing low molecular weight hyaluronic acid higher than high molecular weight hyaluronate acid and vehicle?
2. Is the transepidermal water loss in the elderly after using moisturizers containing high molecular weight hyaluronic acid lower than low molecular weight hyaluronate acid and vehicle?
3. Is the dry skin score (SRRC) in the elderly after using moisturizers containing low molecular weight hyaluronic acid lower than high molecular weight hyaluronate acid and vehicle?
4. Is there any difference in occurence of side effect in elderly between the use of moisturizers containing low molecular weight hyaluronic acid, high molecular weight hyaluronic acid, and vehicle?

ELIGIBILITY:
Inclusion Criteria:

* Female or male diagnosed with xerotic skin
* 60-80 years old
* Willing to participate in clinical trial and sign informed consent

Exclusion Criteria:

* History of hypersensitivity to moisturizer
* Dermatitis or any dermatosis on intervention area in the leg
* Score of erythema and crack more than 2, based on SRRC scoring

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2023-08-26 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Skin capacitance | 2 weeks and 4 weeks
  Skin capacitance is measured by Corneometer CM825
Transepidermal water loss | 2 weeks and 4 weeks
  Transepidermal water loss is measured by Tewameter TM300
Specified symptom sum score/scale, roughness, redness, crack (SRRC) | 2 weeks and 4 weeks
  Evaluation of squama/scale, roughness, redness, and crack of the skin, with a value range of 0-16. Higher values mean worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: Parikesit Muhammad, MD, Principal Investigator — Faculty of Medicine, University of Indonesia
Locations (1):
- Panti Sosial Tresna Werdha Budi Mulia 3, Jakarta, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Pavicic T, Gauglitz GG, Lersch P, Schwach-Abdellaoui K, Malle B, Korting HC, Farwick M. Efficacy of cream-based novel formulations of hyaluronic acid of different molecular weights in anti-wrinkle treatment. J Drugs Dermatol. 2011 Sep;10(9):990-1000. PMID 22052267
- [Result] Ha NG, Lee SH, Lee EH, Chang M, Yoo J, Lee WJ. Safety and efficacy of a new hydrogel based on hyaluronic acid as cosmeceutical for xerosis. J Cosmet Dermatol. 2022 Dec;21(12):6840-6849. doi: 10.1111/jocd.15368. Epub 2022 Sep 20. PMID 36074117
- [Derived] Muhammad P, Novianto E, Setyorini M, Legiawati L, Yusharyahya SN, Menaldi SL, Budianti WK. Effectiveness of topical hyaluronic acid of different molecular weights in xerosis cutis treatment in elderly: a double-blind, randomized controlled trial. Arch Dermatol Res. 2024 Jun 3;316(6):329. doi: 10.1007/s00403-024-03003-2. PMID 38829483